CLINICAL TRIAL: NCT01666340
Title: Generation 100: How Exercise Affects Mortality and Morbidity in the Elderly: A Randomized Control Study
Acronym: GEN100
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Generation-100
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Ageing
Keywords: Exercise; Elderly; Mortality; Morbidity; Prognosis; Longevity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity aerobic training (Experimental): Exercise intervention: High intensity group performing high intensity training where they are required to raise their heart rate several times during the workout and reach perceived exhaustion of 16 on a Borg scale
  Interventions: Other: Exercise intervention
- Moderate intensity training (Other): Exercise intervention: Moderate intensity Group of people asked to perform moderate training where they exercise at a given intensity (moderate as per Borg scale) for a certain amount of time
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — Group asked to perform exercise at a given moderate intensity for a set time
  Other Names: Moderate training
Other: Exercise intervention — High intensity exercise
  Other Names: High intensity

SUMMARY:
Hypothesis: Exercise will reduce morbidity and mortality rates in an elderly population. The extent of reduction will be intensity dependent.

DETAILED DESCRIPTION:
Literature lacks large controlled randomized studies that look at the effect of exercise training on morbidity and mortality. Generation 100 will be the first randomized, controlled clinical study where the primary objective is to study the effects of exercise training on morbidity and mortality in the elderly. Furthermore, the researchers will investigate whether there is a relationship between the exercise intensity and health benefits, with particular focus on major health problems in the elderly population. In addition to being a study, this is also an initiative to improve public health in all healthy individuals between 70-75 years of age in the Trondheim municipality. The participants will either be randomized to supervised exercise or follow current guidelines for physical activity on their own. Clinical examinations, as well as questionnaires, will be administered to all participants at baseline, after one year, after three years, and after five years. Additionally, participants will be followed-up by linking to relevant registers for up to 20 years.

Also data will be collected with the purposes of (a) investigating genetic predisposition for fitness and cardiovascular diseases, and (b) identification of potential targets for therapies.

The study seeks to determine if exercise training gives the seniors a longer active and healthy life.

ELIGIBILITY:
Inclusion Criteria:

* Born in 1936, 1937, 1938, 1939, 1940, 1941 or 1942
* Able to complete the exercise program (determined by the researchers).

Exclusion Criteria:

* Illness or disabilities that preclude exercise or hinder completion of the study
* Uncontrolled hypertension
* Symptomatic valvular, hypertrophic cardiomyopathy, unstable angina, pulmonary hypertension, heart failure and severe arrhythmia
* Diagnosed dementia
* Cancer that makes participation impossible or exercise contraindicated. Considered individually, in consultation with the attending physician.
* Chronic communicable infectious diseases.
* Test results indicating that study participation is unsafe
* Participation in other studies conflicting with participation in Generation 100

Ages: 70 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1567 (Actual)
Dates: Start 2012-08-21 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years follow up
  using data from governmental registers

SECONDARY OUTCOMES:
General measurements | 1 year follow up, 3 years follow up, 5 years follow up
  resting blood pressure, resting fasting blood sample, resting heart rate, weight, height and waistline, body composition (muscle vs fat) questionnaires (activity, safety, monthly training diary) walking test, grip strength test, leg strength test, pulmonary function, physical activity level
Epigenetics | 1 year follow up, 3 years follow up, 5 years follow up
  transcriptomics (messenger RNAs and microRNAs) and proteomics arrays, aimed at blood-borne factors induced by training.
Morbidity | 3 and 5 years
  Look at morbidity after 3 and 5 years follow up(i.e. cardiovascular disease, cancer, etc.) using medical records and link to the different health registers.
Mortality and Morbidity | 10 years
  Look at morbidity after 10 year follow-up

OTHER OUTCOMES:
Cognitive screening | 1 year follow up, 3 years follow up, 5 years follow ut
  Mini Mental Status (MMS)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, Professor, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Background] Stensvold D, Viken H, Rognmo O, Skogvoll E, Steinshamn S, Vatten LJ, Coombes JS, Anderssen SA, Magnussen J, Ingebrigtsen JE, Fiatarone Singh MA, Langhammer A, Stoylen A, Helbostad JL, Wisloff U. A randomised controlled study of the long-term effects of exercise training on mortality in elderly people: study protocol for the Generation 100 study. BMJ Open. 2015 Feb 12;5(2):e007519. doi: 10.1136/bmjopen-2014-007519. PMID 25678546
- [Background] Viken H, Reitlo LS, Zisko N, Nauman J, Aspvik NP, Ingebrigtsen JE, Wisloff U, Stensvold D. Predictors of Dropout in Exercise Trials in Older Adults: The Generation 100 Study. Med Sci Sports Exerc. 2019 Jan;51(1):49-55. doi: 10.1249/MSS.0000000000001742. PMID 30113524
- [Result] Stensvold D, Viken H, Steinshamn SL, Dalen H, Stoylen A, Loennechen JP, Reitlo LS, Zisko N, Baekkerud FH, Tari AR, Sandbakk SB, Carlsen T, Ingebrigtsen JE, Lydersen S, Mattsson E, Anderssen SA, Fiatarone Singh MA, Coombes JS, Skogvoll E, Vatten LJ, Helbostad JL, Rognmo O, Wisloff U. Effect of exercise training for five years on all cause mortality in older adults-the Generation 100 study: randomised controlled trial. BMJ. 2020 Oct 7;371:m3485. doi: 10.1136/bmj.m3485. PMID 33028588
- [Result] Letnes JM, Berglund I, Johnson KE, Dalen H, Nes BM, Lydersen S, Viken H, Hassel E, Steinshamn S, Vesterbekkmo EK, Stoylen A, Reitlo LS, Zisko N, Baekkerud FH, Tari AR, Ingebrigtsen JE, Sandbakk SB, Carlsen T, Anderssen SA, Singh MAF, Coombes JS, Helbostad JL, Rognmo O, Wisloff U, Stensvold D. Effect of 5 years of exercise training on the cardiovascular risk profile of older adults: the Generation 100 randomized trial. Eur Heart J. 2022 Jun 1;43(21):2065-2075. doi: 10.1093/eurheartj/ehab721. PMID 34746955
- [Derived] Bakken J, Brissach DE, Ingestrom EML, Midttun S, Walker TL, Stensvold D, Tari AR. Effects of 5-Year Exercise Training on Cognition in Older Adults: 10-Years Follow-Up from the Generation 100 Study. Sports Med Open. 2025 Dec 7;11(1):153. doi: 10.1186/s40798-025-00956-0. PMID 41354893
- [Derived] Hallan SI, Ovrehus MA, Shlipak MG, Potok OA, Romundstad S, Aspvik NP, Wisloff U, Ix JH, Stensvold D, Langlo KA. Long-Term Physical Exercise for Preventing CKD in Older Adults: A Randomized Clinical Trial. J Am Soc Nephrol. 2025 Feb 11;36(7):1352-1362. doi: 10.1681/ASN.0000000636. PMID 39932787
- [Derived] Tari AR, Brissach DE, Ingestrom EML, Nauman J, Tyrell T, Foster C, Radtke K, Porcari JP, Lydersen S, Kaminsky LA, Myers J, Walker TL, Coombes JS, Stensvold D, Wisloff U. Survival of the fittest? Peak oxygen uptake and all-cause mortality among older adults in Norway. Prog Cardiovasc Dis. 2025 Mar-Apr;89:25-34. doi: 10.1016/j.pcad.2024.11.004. Epub 2024 Dec 4. PMID 39638222
- [Derived] Reitlo LS, Mihailovic JM, Stensvold D, Wisloff U, Hyder F, Haberg AK. Hippocampal neurochemicals are associated with exercise group and intensity, psychological health, and general cognition in older adults. Geroscience. 2023 Jun;45(3):1667-1685. doi: 10.1007/s11357-022-00719-9. Epub 2023 Jan 10. PMID 36626020
- [Derived] Zotcheva E, Haberg AK, Wisloff U, Salvesen O, Selbaek G, Stensvold D, Ernstsen L. Effects of 5 Years Aerobic Exercise on Cognition in Older Adults: The Generation 100 Study: A Randomized Controlled Trial. Sports Med. 2022 Jul;52(7):1689-1699. doi: 10.1007/s40279-021-01608-5. Epub 2021 Dec 8. PMID 34878637
- [Derived] Sokolowski DR, Hansen TI, Rise HH, Reitlo LS, Wisloff U, Stensvold D, Haberg AK. 5 Years of Exercise Intervention Did Not Benefit Cognition Compared to the Physical Activity Guidelines in Older Adults, but Higher Cardiorespiratory Fitness Did. A Generation 100 Substudy. Front Aging Neurosci. 2021 Nov 16;13:742587. doi: 10.3389/fnagi.2021.742587. eCollection 2021. PMID 34867275
- [Derived] Berglund I, Vesterbekkmo EK, Retterstol K, Anderssen SA, Fiatarone Singh MA, Helge JW, Lydersen S, Wisloff U, Stensvold D. The Long-term Effect of Different Exercise Intensities on High-Density Lipoprotein Cholesterol in Older Men and Women Using the Per Protocol Approach: The Generation 100 Study. Mayo Clin Proc Innov Qual Outcomes. 2021 Sep 16;5(5):859-871. doi: 10.1016/j.mayocpiqo.2021.07.002. eCollection 2021 Oct. PMID 34585083
- See also: Generation 100 web page — http://www.ntnu.edu/cerg/generation100
- See also: Results published in BMJ Oct 2020 — https://doi.org/10.1136/bmj.m3485